CLINICAL TRIAL: NCT02361281
Title: Validation of a Previously Performed Study on Non-invasive Diagnostic Method for Sarcoidosis Using Exhaled Breath
Brief Title: Validation of a Non-invasive Diagnostic Method for Sarcoidosis Using Exhaled Breath
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Maastricht University (Other)
Collaborators: Gelderse Vallei Hospital (Other); Atrium Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: BC/1408-389
Record Dates: First submitted 2015-02-02; First posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sarcoidosis patients: Clinically relevant sarcoidosis patients with different stages and treatments.
- Healthy controls: Healthy people without any pulmonary conditions

SUMMARY:
Sarcoidosis is a chronic lung disease that is characterized by fatigue, shortness of breath, chest pain and reduced lung function. Suffering from these diseases has a very negative effect on the quality of life. When people are suspected of having sarcoidosis various markers in the blood are measured. Ultimate diagnosis, however, always requires invasive techniques such as bronchoscopy and lung biopsy. Consequently, there is an urgent need for a new diagnostic tool that is easy, quick and most of all non-invasive and thus friendly for the patient.

Such a new diagnostic tool might be found in examining the exhaled air of patients, which contains a complex mixture of so-called volatile organic compounds (VOCs) that are the result of damaging processes that occur in the lung. Determining the VOC profile in the breath can be used as a biomarker, or biological indicator, of those damaging processes. In other words, searching for unique VOC profiles in the breath of sarcoidosis patients might lead to the development of a diagnostic tool that only uses their exhaled breath.

The current study involves 25 sarcoidosis patients and 25 healthy volunteers. The aim of this study is find VOCs in exhaled air that can be used to diagnose sarcoidosis. In a previous study, sarcoidosis-specific VOCs were found, which we intend to validate using the current study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed sarcoidosis

Exclusion Criteria:

* (ex-) smokers
* for healthy controls: controls with pulmonary disease excluded

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: sarcoidosis patients with confirmed disease, with a range of disease stages. Average age for all study subjects: +- 50 y/o male/female ratio: approx 15 men vs. 10 women in each group.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-03 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
diagnosis by exhaled breath | upon regular visit to clinic, which is expected to occur on average within 4 months after the start of the study

CONTACTS AND LOCATIONS:
Overall Officials: Rianne Fijten, MSc, Principal Investigator — Maastricht University

REFERENCES:
- [Derived] Fijten RRR, Smolinska A, Drent M, Dallinga JW, Mostard R, Pachen DM, van Schooten FJ, Boots AW. The necessity of external validation in exhaled breath research: a case study of sarcoidosis. J Breath Res. 2017 Nov 29;12(1):016004. doi: 10.1088/1752-7163/aa8409. PMID 28775245